CLINICAL TRIAL: NCT05732142
Title: Postpartum Integration of Vaccines and Contraception Trial
Acronym: PIVoT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 804819
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Contraception; Gender Equity
Keywords: Family Planning; Infant Vaccination; Linked Care; India

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PIVoT (Experimental): Gender-transformative family planning counseling and contraception provision at the time of infant vaccination
  Interventions: Other: Postpartum Integration of Vaccines and Contraception Through Gender-Transformative Programming(PIVoT)
- Standard of care (No Intervention): Standard infant vaccination and family planning referrals

INTERVENTIONS:
Other: Postpartum Integration of Vaccines and Contraception Through Gender-Transformative Programming(PIVoT) — The PIVoT intervention is a 30-minute focused information exchange that supports shared contraceptive decision making. The program includes a gender-equity and family planning curriculum covering basic family planning information as well as gender norms and son preference and interactive family planning method index cards (detailing method characteristics, use, duration of action, efficacy, side effects, and contraindications for each method). The program is designed to support person-centered contraceptive choice and encourages women to consider joint family planning decision-making with male partners. If a contraceptive method is desired, it will be provided by nurses who are trained to provide comprehensive family planning care.
  Arms: PIVoT

SUMMARY:
This study aims to examine how to implement a gender-transformative post-partum family planning program integrated into community-based infant vaccination services, and to evaluate preliminary effectiveness of this approach on postpartum contraceptive use in a low resource, rural setting.

DETAILED DESCRIPTION:
Using effective postpartum contraception allows postpartum people to prevent short inter-pregnancy intervals which are associated with an increased risk of maternal and infant morbidity and mortality. India is the country with the highest number of women with an unmet need for contraception, and postpartum and rural women are those with the greatest need. Uptake of postpartum contraception among women in rural India is low; less than half of postpartum women use contraception within the first year after delivery, and many births do not follow the recommended interval.

A promising intervention to address barriers to family planning care is to build on an existing successful health program, the infant vaccination program, by linking family planning services with infant vaccination. India's Ministry of Health has promoted community-based delivery of infant vaccinations, and monthly childhood vaccination services are offered at Village Health and Nutrition Days typically held at Anganwadi Community Centers. Six-week vaccination rates are high, indicating that these services are routinely used by families of young infants, which provides an opportunity to reach postpartum women simultaneously. This programming addresses gender-inequitable social norms and has shown to facilitate more successful family planning intervention but has not been studied among postpartum women. This study will adapt a gender-transformative family planning intervention to support community-based delivery of family planning with infant vaccination; this intervention has the potential to increase family planning use among postpartum women with unmet need in low-resources and rural settings.

This is a two-arm, cluster randomized-trial where postpartum women will be assigned to participation in the linked care model (PIVoT) or the standard of care (referring women to public health centers for family planning counseling and contraceptive provision). The study team will enroll 286 women in the study, 143 in each the intervention and control arms. Randomization will occur at the subcenter level. Participants will be recruited among postpartum women presenting for infant vaccination services at VHND.

Follow-up will occur with women at 6 months and 12 months postpartum and outcomes will be assessed via tablet-based surveys. In addition, a total of 40 in-depth interviews will take place with a group of PIVoT intervention participants, their husbands, and health care providers who delivered the program after completion of the study for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who delivered a baby within the past 12 weeks
* Speak Marathi
* Reside in rural Maharashtra
* Did not undergo sterilization, hysterectomy or immediate postpartum intrauterine device (IUD) placement

Exclusion Criteria:

* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women using modern contraception at 6 months postpartum | 6 months after delivery
  Contraceptive use will be measured through a self-reported survey collected at 6 months postpartum.

SECONDARY OUTCOMES:
Feasibility, acceptability and appropriateness of the PiVOT intervention (quantitative) | 6 months after delivery
  Self-reported survey questions using validated items regarding feasibility, acceptability and appropriateness of linked care will be collected at 6 months postpartum. Participants will rate the 3 constructs using 12 items comprising 3 4-item scales with a 5-point Likert scale: completely agree=1, agree=2, neither agree nor disagree=3, disagree=4, completely disagree=5. Higher scores on these items reflect more supportive attitudes toward the linked care model.
Proportion of women using modern contraception at 12 months postpartum | 12 months after delivery
  Contraceptive use will be measured through a self-reported survey collected at 12 months postpartum
Feasibility, acceptability and appropriateness of the PiVOT intervention (qualitative) among participants | 6 months postpartum
  In-depth interviews with a portion of PiVOT intervention participants
Feasibility, acceptability and appropriateness of the PiVOT intervention (qualitative) among providers of the program | 6 months postpartum
  In-depth interviews with health care providers who delivered the PIVoT intervention after completion of the research study to further understand this outcome using qualitative data.
Feasibility, acceptability and appropriateness of the PiVOT intervention (qualitative) among husbands of participants | 6 months postpartum
  In-depth interviews with husbands of participants (if recommended by their wife) after completion of the research study to further understand this outcome using qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, MAS, Principal Investigator — University of California, San Diego; Shahina Begum, PhD, Principal Investigator — Indian Council of Medical Research-National Institute for Research in Reproductive and Child Health
Locations (2):
- University of California, San Diego, La Jolla, California, United States
- Junnar Taluka, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No